CLINICAL TRIAL: NCT02480751
Title: TRK-100STP PhaseII Clinical Study -Chronic Renal Failure (Primary Glomerular Disease/Nephrosclerosis)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100CRS01/533-CL-00
Record Dates: First submitted 2015-06-21; First posted 2015-06-24 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Chronic Renal Failure; Prostaglandin; Prostacyclin; Glomerular Disease; Nephrosclerosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Nephrosclerosis | interventions — beraprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1: Exprimental (TRK-100STP) (Experimental): high dose
  Interventions: Drug: Beraprost
- 2: Exprimental (TRK-100STP) (Experimental): low dose
  Interventions: Drug: Beraprost
- 3: Placebo Comparator (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Beraprost
  Arms: 1: Exprimental (TRK-100STP); 2: Exprimental (TRK-100STP)
Drug: Placebo
  Arms: 3: Placebo Comparator

SUMMARY:
The purpose of this study is to determine the recommended dose of the sustained-release form of BPS (TRK-100STP low dose or high dose) in Japanese patients with CRF (Primary glomerular disease/nephrosclerosis).

ELIGIBILITY:
Inclusion Criteria:

* The CRF patient with primary glomerular disease or nephrosclerosis as the primary disease
* The patient with progressive CRF

Exclusion Criteria:

* The patient with secondary glomerular disease
* The patient with CRF caused by pyelonephritis, interstitial/tubular nephritis, gouty kidney, polycystic kidney disease, or nephroureterolithiasis

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Difference between the run-in and treatment periods in the slope of the regression line of 1/SCr versus time | 50 weeks (Run-in 22weeks, Treatment 28 weeks)

REFERENCES:
- [Derived] Koyama A, Fujita T, Gejyo F, Origasa H, Isono M, Kurumatani H, Okada K, Kanoh H, Kiriyama T, Yamada S. Orally active prostacyclin analogue beraprost sodium in patients with chronic kidney disease: a randomized, double-blind, placebo-controlled, phase II dose finding trial. BMC Nephrol. 2015 Oct 16;16:165. doi: 10.1186/s12882-015-0130-5. PMID 26475266